CLINICAL TRIAL: NCT00345930
Title: A Multi-Center, Longitudinal Study of Drug-and CAM-Induced Liver Injury
Brief Title: DILIN - Prospective Study
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00113362_1; U01DK065176 (NIH); Pro00072297 (Other: Advarra); Pro00017208 (Other: Original Duke IRB number)
Record Dates: First submitted 2006-06-27; First posted 2006-06-29 (Estimated); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Liver Diseases
Keywords: Complementary and alternative medicine; Complementary therapies; Alternative therapies; Prescription Drugs; Non prescription Drugs; Liver Disease; Chemical Ind; Phenotype; Proteomics; Metabolomics; Cholestatic Liver Injury; Hepatocellular Liver Injury; Mixed Liver Injury; Matched Case Control Studies; Genotype; Liver Dis; Chem Ind
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2: Individuals without drug induced liver disease
- 1: Individuals with drug induced liver disease

SUMMARY:
The purpose of this study is to identify individuals who have suffered a liver injury arising as an idiosyncratic reaction to a prescription drug or a complementary and alternative medicine. Recently added acute cases enrollment that meets criteria to the protocol. Also added Fibroscans to the protocol that will be completed at baseline and follow-up on chronic subjects.

DETAILED DESCRIPTION:
Liver injury due to prescription and non-prescription medication use is a medical, scientific and public health problem of increasing frequency and importance in the United States. Indeed, drug-induced liver injury (DILI) is the most important reason for non-approval, withdrawal, limitation in use and clinical monitoring by the Food and Drug Administration (FDA). However, detection of signals for liver injury frequently relies upon the reporting of cases by practitioners to health authorities in post-marketing surveillance. Under-reporting of cases, lack of mandatory reporting systems, and difficulties in establishing a diagnosis make the current system sub-optimal. Moreover, with the growing use of complementary and alternative medications (CAM), there have also been increasing reports of liver toxicity due to various non-prescription herbal, dietary and food additive supplements. Because the manufacturing, dispensing and testing of these products is not regulated, the hepatotoxic potential of these formulations is poorly characterized or completely unknown.

The DILIN Prospective Study is a multi-centered epidemiological study designed to gather clinical information and biological specimens on cases of suspected liver injury due to drugs and CAM. The goals of this study are to develop a database of recent DILI cases, identify the clinical, environmental and genetic risk factors that predict DILI, develop standardized instruments and terminology and perform careful longitudinal follow-up of DILI subjects. Biological samples collected will be used in future studies of the mechanisms and genetics of DILI.

Patients who are referred to one of the DILIN clinical sites and who, in the opinion of gastroenterologist/hepatologist, experienced a drug-induced liver injury are enrolled. Detailed clinical data and biological specimens are collected. Clinical data will be reviewed by the DILIN Causality Committee and the final determination on whether the subject qualifies as a bona fide DILI case is made by consensus opinion. DILI cases (only) are followed for at least 6 months to derive the longitudinal profile of drug-and CAM-induced liver injury. Detailed clinical data including liver elastography (FibroScans) and biological specimens are collected. Patients who satisfy the definition of chronic DILI will be evaluated with additional FibroScans at 12, 24, 36 and 48 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Age > 2 years at enrollment into the study.
* Evidence of liver injury that is known or suspected to be related to consumption of a drug or CAM product in the 6-month period prior to enrollment.
* Written Informed consent from the patient or the patient's legal guardian.
* Documented clinically important DILI, defined as any of the following:

  1. ALT or AST >5 x ULN or A P'ase >2 x ULN confirmed on at least 2 consecutive blood draws in patients with previously normal values.
  2. If baseline (BL) ALT, AST or A P'ase are known to be elevated, then ALT or AST >5 x BL or A P'ase >2 x BL on at least 2 consecutive blood draws. "Baseline" is defined as the average of at least 2 measurements performed during the 12-month period prior to starting the DILI medication.
  3. Any elevation of ALT, A P'ase, or AST, associated with (a) increased total bilirubin [ ≥ 2.5 mg/dL], in absence of prior diagnosis of liver disease, Gilbert's syndrome, or evidence of hemolysis or (b) coagulopathy with INR > 1.5 in absence of coumadin therapy or known vitamin K deficiency.

Exclusion Criteria:

Patients with any of the following will not be eligible for participation:

* Competing cause of acute liver injury such as hepatic ischemia that is felt by the investigator to be the primary reason for observed liver injury and supported by laboratory tests, serologies, liver biopsy, or radiology.
* Known, pre-existing autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, or other chronic biliary tract disease which may confound the ability to make a diagnosis of DILI.
* Acetaminophen hepatotoxicity.
* Liver/bone marrow transplant prior to the development of drug- or CAM-induced liver injury.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have suffered a drug induced liver injury and meet inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2004-09 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Develop a database of recent DILI cases | July 2028
  develop a database of recent DILI cases

CONTACTS AND LOCATIONS:
Overall Officials: Huiman X. Barnhart, PhD, Principal Investigator — Duke University; Robert Fontana, MD, Study Chair — Univ. of Michiganl
Locations (6):
- United States (6):
  - University of Southern California, Los Angeles, California
  - Indiana University, Indianapolis, Indiana
  - NIH Clinical Site, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Univeristy of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Thomas Jefferson, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Fontana RJ, Watkins PB, Bonkovsky HL, Chalasani N, Davern T, Serrano J, Rochon J; DILIN Study Group. Drug-Induced Liver Injury Network (DILIN) prospective study: rationale, design and conduct. Drug Saf. 2009;32(1):55-68. doi: 10.2165/00002018-200932010-00005. PMID 19132805
- [Background] Chalasani N, Fontana RJ, Bonkovsky HL, Watkins PB, Davern T, Serrano J, Yang H, Rochon J; Drug Induced Liver Injury Network (DILIN). Causes, clinical features, and outcomes from a prospective study of drug-induced liver injury in the United States. Gastroenterology. 2008 Dec;135(6):1924-34, 1934.e1-4. doi: 10.1053/j.gastro.2008.09.011. Epub 2008 Sep 17. PMID 18955056
- [Derived] Gopalakrishna H, Ghabril M, Gu J, Li YJ, Fontana RJ, Kleiner DE, Koh C, Chalasani N; Drug-Induced Liver Injury Network. Drug-induced Liver Injury Due to Medications for Alcohol Use Disorder: Results From the DILIN Prospective Study. J Addict Med. 2025 May-Jun 01;19(3):314-321. doi: 10.1097/ADM.0000000000001421. Epub 2024 Dec 9. PMID 39651750
- [Derived] Fontana RJ, Kleiner DE, Chalasani N, Bonkovsky H, Gu J, Barnhart H, Li YJ, Hoofnagle JH. The Impact of Patient Age and Corticosteroids in Patients With Sulfonamide Hepatotoxicity. Am J Gastroenterol. 2023 Sep 1;118(9):1566-1575. doi: 10.14309/ajg.0000000000002232. Epub 2023 Feb 27. PMID 36848311
- [Derived] Fontana RJ, Engle RE, Hayashi PH, Gu J, Kleiner DE, Nguyen H, Barnhart H, Hoofnagle JH, Farci P. Incidence of Hepatitis E Infection in American Patients With Suspected Drug-Induced Liver Injury Is Low and Declining: The DILIN Prospective Study. Am J Gastroenterol. 2022 Sep 1;117(9):1462-1470. doi: 10.14309/ajg.0000000000001869. Epub 2022 Jun 10. PMID 35973149
- [Derived] Devarbhavi H, Ghabril M, Barnhart H, Patil M, Raj S, Gu J, Chalasani N, Bonkovsky HL. Leflunomide-induced liver injury: Differences in characteristics and outcomes in Indian and US registries. Liver Int. 2022 Jun;42(6):1323-1329. doi: 10.1111/liv.15189. Epub 2022 Feb 15. PMID 35129282
- [Derived] Vuppalanchi R, Bonkovsky HL, Ahmad J, Barnhart H, Durazo F, Fontana RJ, Gu J, Khan I, Kleiner DE, Koh C, Rockey DC, Phillips EJ, Li YJ, Serrano J, Stolz A, Tillmann HL, Seeff LB, Hoofnagle JH, Navarro VJ; Drug-Induced Liver Injury Network. Garcinia cambogia, Either Alone or in Combination With Green Tea, Causes Moderate to Severe Liver Injury. Clin Gastroenterol Hepatol. 2022 Jun;20(6):e1416-e1425. doi: 10.1016/j.cgh.2021.08.015. Epub 2021 Aug 14. PMID 34400337
- [Derived] Martinez MA, Vuppalanchi R, Fontana RJ, Stolz A, Kleiner DE, Hayashi PH, Gu J, Hoofnagle JH, Chalasani N. Clinical and histologic features of azithromycin-induced liver injury. Clin Gastroenterol Hepatol. 2015 Feb;13(2):369-376.e3. doi: 10.1016/j.cgh.2014.07.054. Epub 2014 Aug 9. PMID 25111234
- [Derived] Navarro VJ, Barnhart H, Bonkovsky HL, Davern T, Fontana RJ, Grant L, Reddy KR, Seeff LB, Serrano J, Sherker AH, Stolz A, Talwalkar J, Vega M, Vuppalanchi R. Liver injury from herbals and dietary supplements in the U.S. Drug-Induced Liver Injury Network. Hepatology. 2014 Oct;60(4):1399-408. doi: 10.1002/hep.27317. Epub 2014 Aug 25. PMID 25043597
- [Derived] Ghabril M, Bonkovsky HL, Kum C, Davern T, Hayashi PH, Kleiner DE, Serrano J, Rochon J, Fontana RJ, Bonacini M; US Drug-Induced Liver Injury Network. Liver injury from tumor necrosis factor-alpha antagonists: analysis of thirty-four cases. Clin Gastroenterol Hepatol. 2013 May;11(5):558-564.e3. doi: 10.1016/j.cgh.2012.12.025. Epub 2013 Jan 17. PMID 23333219
- See also: Multi-center, Longitudinal Study of Drug- and CAM-Induced Liver Injury. — https://dilin.org/
- See also: The National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) conducts and supports biomedical research and disseminates research findings & health information to the public. — http://www.niddk.nih.gov